CLINICAL TRIAL: NCT00068250
Title: Phase I/II Study Of Pre-Irradiation Chemotherapy With Methotrexate, Rituximab, And Temozolomide And Post -Irradiation Temozolomide For Primary Central Nervous System Lymphoma
Brief Title: Combination Chemotherapy, Monoclonal Antibody, and Radiation Therapy in Treating Patients With Primary Central Nervous System Lymphoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Radiation Therapy Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH); NRG Oncology (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: RTOG-0227; CDR0000301563
Record Dates: First submitted 2003-09-10; First posted 2003-09-11 (Estimated); Results first posted 2018-02-07 (Actual); Last update posted 2018-02-07 (Actual); Status verified 2018-02

CONDITIONS: Brain and Central Nervous System Tumors; Lymphoma
Keywords: primary central nervous system non-Hodgkin lymphoma; primary central nervous system Hodgkin lymphoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Lymphoma | interventions — Rituximab; Methotrexate; Temozolomide; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Phase I: Temozolomide 100 mg (Experimental): Rituximab, methotrexate, temozolomide 100 mg/m^2, followed by radiation therapy, then post-radiation therapy temozolomide 200 mg/m^2.
  Interventions: Drug: rituximab; Drug: methotrexate; Drug: temozolomide 100 mg/m^2; Radiation: radiation therapy; Drug: post-radiation therapy temozolomide
- Phase I: Temozolomide 150 mg (Experimental): Rituximab, methotrexate, temozolomide 150 mg/m^2, followed by radiation therapy, then post-radiation therapy temozolomide 200 mg/m^2.
  Interventions: Drug: rituximab; Drug: methotrexate; Drug: temozolomide 150 mg/m^2; Radiation: radiation therapy; Drug: post-radiation therapy temozolomide
- Phase I: Temozolomide 200 mg (Experimental): Rituximab, methotrexate, temozolomide 200 mg/m^2, followed by radiation therapy, then post-radiation therapy temozolomide 200 mg/m^2.
  Interventions: Drug: rituximab; Drug: methotrexate; Drug: temozolomide 200 mg/m^2; Radiation: radiation therapy; Drug: post-radiation therapy temozolomide
- Phase II: Temozolomide 100 mg (Experimental): Rituximab, methotrexate, temozolomide 100 mg/m^2, followed by radiation therapy, then post-radiation therapy temozolomide 200 mg/m^2.
  Interventions: Drug: rituximab; Drug: methotrexate; Drug: temozolomide 100 mg/m^2; Radiation: radiation therapy; Drug: post-radiation therapy temozolomide

INTERVENTIONS:
Drug: rituximab — 375 mg/m2, intravenously three days prior to the first cycle of methotrexate
Drug: methotrexate — Five cycles of methotrexate (MTX) at 3.5 gm/m2 administered every two weeks on weeks 1, 3, 5, 7, and 9 via intravenous infusion over four hours once per cycle. Calcium leucovorin 25 mg orally or intravenously every six hours initiated exactly 24 hours following the start of the MTX infusion. Methotrexate levels to be monitored daily, and calcium leucovorin discontinued when the MTX level is less than 10 micromolar.
Drug: temozolomide 100 mg/m^2 — Temozolomide 100 mg/m^2 by mouth per day for five days on weeks 4 and 8.
  Arms: Phase I: Temozolomide 100 mg; Phase II: Temozolomide 100 mg
Drug: temozolomide 150 mg/m^2 — Temozolomide 150 mg/m^2 by mouth per day for five days on weeks 4 and 8.
  Arms: Phase I: Temozolomide 150 mg
Drug: temozolomide 200 mg/m^2 — Temozolomide 200 mg/m^2 per day by mouth for five days on weeks 4 and 8.
  Arms: Phase I: Temozolomide 200 mg
Radiation: radiation therapy — Whole brain irradiation (WBRT) during weeks 11, 12, and 13, five days per week (excluding weekends). A daily dose of 2.4 Gy delivered in two fractions of 1.2 Gy each with a minimum inter-fraction interval of 6 hours, with a total dose to brain and meninges of 36 Gy.
  Other Names: radiotherapy
Drug: post-radiation therapy temozolomide — Temozolomide (TMZ) 200 mg/m^2 by mouth per day for 5 days on weeks 14, 18, 22, 26, 30, 34, 38, 42, 46, and 50 for a total of 10 cycles.

SUMMARY:
RATIONALE: Drugs used in chemotherapy such as methotrexate and temozolomide use different ways to stop cancer cells from dividing so they stop growing or die. Monoclonal antibodies such as rituximab can locate cancer cells and either kill them or deliver cancer-killing substances to them without harming normal cells. Radiation therapy uses high-energy x-rays to damage cancer cells. Combining methotrexate, temozolomide, and rituximab with radiation therapy may kill more cancer cells.

PURPOSE: This phase I/II trial is studying the side effects and best dose of temozolomide when given together with methotrexate and rituximab followed by radiation therapy and to see how well they work in treating patients with primary central nervous system lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* To assess the maximum tolerated dose (MTD) of temozolomide (TMZ) in combination with methotrexate (MTX) and rituximab (RTX) when administered prior to twice daily fractionated whole brain radiation therapy (WBRT) in patients with primary central nervous system lymphoma.
* To compare the two-year survival rate in patients receiving pre-irradiation chemotherapy, twice daily fractionated whole brain radiation therapy and post-irradiation temozolomide to the reported two-year survival rate of Radiation Therapy Oncology Group (RTOG) trial 93-10. RTOG 9310 does not fall within ClinicalTrials.gov registration/reporting requirements.)
* To compare the pre-irradiation chemotherapy tumor response rates to the reported rate from RTOG 93-10.
* To report progression-free survival.
* To assess acute and long-term neurologic toxicity, and to collect quality of life data for this patient group.

Patients are followed every 3 months for 2 years, every 6 months for 3 years, and then annually thereafter.

ELIGIBILITY:
Inclusion criteria:

1. Primary central nervous system (CNS) lymphoma [B-cell, Cluster of Differentiation 20 (CD20) antigen positive] based on positive biopsy or cerebrospinal fluid (CSF) or vitreous cytology (in association with measurable intraparenchymal tumor). Cytology must demonstrate lymphoma or have an immunohistochemical diagnosis of malignant lymphocytes with a monoclonal lymphocytic population.
2. Life expectancy ≥ 8 weeks;
3. Zubrod performance status of 0-2;
4. Absolute granulocyte count ≥1500/mm3; platelet count ≥ 100,000/mm3; creatinine clearance ≥ 50, calculated with the Cockcroft-Gault Equation: Cr Clearance = (140-age) x wt (kg)/(Cr[mg/dl]x 72); Bilirubin, serum glutamate oxaloacetate transaminase (SGOT), alkaline phosphatase (AST) ≤ 2 x institutional upper limits of normal;
5. Patients must sign a study-specific informed consent prior to study entry.
6. Age ≥ 18

Exclusion criteria:

1. Evidence of systemic lymphoma;
2. Prior malignancy (excluding in situ carcinoma of the cervix or non-melanomatous skin cancer)unless disease free for at least five years;
3. Prior radiotherapy to the brain or head/neck;
4. Prior chemotherapy;
5. History of idiopathic sensitivity to any of the drugs to be used;
6. Active infectious process;
7. Seropositive for HIV, AIDS, or post-organ transplant;
8. Pregnant women are ineligible as treatment involves unforeseeable risks to the participant and to the embryo or fetus.
9. Active hepatitis B.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2003-07; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jon Glass, MD, Study Chair — Sidney Kimmel Cancer Center at Thomas Jefferson University
Locations (26):
- United States (26):
  - Baptist Cancer Institute - Jacksonville, Jacksonville, Florida
  - Integrated Community Oncology Network at Southside Cancer Center, Jacksonville, Florida
  - Baptist Medical Center South, Jacksonville, Florida
  - Integrated Community Oncology Network, Jacksonville Beach, Florida
  - Integrated Community Oncology Network - Orange Park, Orange Park, Florida
  - Florida Cancer Center - Palatka, Palatka, Florida
  - Flagler Cancer Center, Saint Augustine, Florida
  - Borgess Medical Center, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - CCOP - Kansas City, Kansas City, Missouri
  - Siteman Cancer Center at Barnes-Jewish Hospital - Saint Louis, St Louis, Missouri
  - CCOP - Nevada Cancer Research Foundation, Las Vegas, Nevada
  - John F. Kennedy Medical Center, Edison, New Jersey
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Providence Milwaukie Hospital, Milwaukie, Oregon
  - Providence Cancer Center at Providence Portland Medical Center, Portland, Oregon
  - CCOP - Columbia River Oncology Program, Portland, Oregon
  - Providence St. Vincent Medical Center, Portland, Oregon
  - Kimmel Cancer Center at Thomas Jefferson University - Philadelphia, Philadelphia, Pennsylvania
  - Hollings Cancer Center at Medical University of South Carolina, Charleston, South Carolina
  - Jon and Karen Huntsman Cancer Center at Intermountain Medical Center, Murray, Utah
  - Utah Valley Regional Medical Center - Provo, Provo, Utah
  - Southwest Washington Medical Center Cancer Center, Vancouver, Washington
  - Community Memorial Hospital Cancer Care Center, Menomonee Falls, Wisconsin
  - Medical College of Wisconsin Cancer Center, Milwaukee, Wisconsin

REFERENCES:
- [Result] Glass J, Won M, Schultz CJ, Brat D, Bartlett NL, Suh JH, Werner-Wasik M, Fisher BJ, Liepman MK, Augspurger M, Bokstein F, Bovi JA, Solhjem MC, Mehta MP. Phase I and II Study of Induction Chemotherapy With Methotrexate, Rituximab, and Temozolomide, Followed By Whole-Brain Radiotherapy and Postirradiation Temozolomide for Primary CNS Lymphoma: NRG Oncology RTOG 0227. J Clin Oncol. 2016 May 10;34(14):1620-5. doi: 10.1200/JCO.2015.64.8634. Epub 2016 Mar 28. PMID 27022122

RESULTS

PARTICIPANT FLOW:
Period: Phase I: Dose Level 1
Arm/Group | Phase I: Temozolomide 100 mg | Phase I: Temozolomide 150 mg | Phase I: Temozolomide 200 mg | Phase II: Temozolomide 100 mg
Started | 6 | 0 | 0 | 0
Completed | 6 (Subjects with data available for the primary analysis are considered to have completed the study.) | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0
Period: Phase I: Dose Level 2
Arm/Group | Phase I: Temozolomide 100 mg | Phase I: Temozolomide 150 mg | Phase I: Temozolomide 200 mg | Phase II: Temozolomide 100 mg
Started | 0 | 7 | 0 | 0
Completed | 0 | 6 (Subjects with data available for the primary analysis are considered to have completed the study.) | 0 | 0
Not Completed | 0 | 1 | 0 | 0
Not completed — Protocol Violation | 0 | 1 | 0 | 0
Period: Phase II: Dose Level 2
Arm/Group | Phase I: Temozolomide 100 mg | Phase I: Temozolomide 150 mg | Phase I: Temozolomide 200 mg | Phase II: Temozolomide 100 mg
Started | 0 | 0 | 0 | 47
Completed | 0 | 0 | 0 | 47 (Subjects with data available for the primary analysis are considered to have completed the study.)
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Eligible patients who started study treatment
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase I: Temozolomide 100 mg | Phase I: Temozolomide 150 mg | Phase II: Temozolomide 100 mg | Total
Number analyzed (Participants) | 6 | 6 | 47 | 59
Age, Continuous [Median (Full Range); unit: years] | 57 [43 to 70] | 62 [47 to 72] | 57 [24 to 73] | 57 [24 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 | 24 | 30
  Male | 2 | 4 | 23 | 29

OUTCOME MEASURES:

1. Primary Outcome: Number of Phase I Participants Experiencing Toxicity
Description: A dose limiting toxicity (DLT) is defined as any grade 3 or 4 non-hematological toxicity (other than grade 3 nausea/vomiting) or any hematological toxicity resulting in the discontinuation of temozolomide. Toxicity evaluation for this dose escalation includes all toxicities occurring prior to the start of radiation therapy. If the patient did not receive radiation therapy, then toxicity evaluation included all toxicities occurring through week 15. Any grade 5 toxicity would result in immediate suspension of accrual.
Time Frame: From start of treatment to 10 weeks if radiation therapy received, to 15 weeks if not.
Population: Eligible patients on Phase I arms who started study treatment
Measure: Count of Participants; unit: Participants
Groups:
- Phase I: Temozolomide 100mg: Phase I: Temozolomide 100mg
- Phase I: Temozolomide150 mg: Phase I: Temozolomide 150 mg
Arm/Group | Phase I: Temozolomide 100mg | Phase I: Temozolomide150 mg
Number analyzed (Participants) | 6 | 6
Participants | 1 | 3
Statistical Analysis 1: Comparison: Phase I: Temozolomide 100mg vs Phase I: Temozolomide150 mg; Test type: Other; Dose escalation followed the standard 3+3 design, although up to six patients could be accrued per dose level before suspending accrual for toxicity evaluation. If none of the first three patients (0/3), or one of the first three and none of the second three (1/3 and 0/3), experience a DLT, then the current dose level would be considered acceptable, and the next dose opened. Otherwise, the current dose level would be considered too toxic. The highest dose achieved with an acceptable level of toxicity was to considered the Maximum Tolerable Dose (MTD). If at any time a grade 5 toxicity was observed, accrual will be suspended, and the Study Chair would review the event. Furthermore, if the cumulative incidence (obtained by time to event analysis), at any time, of combined acute/late DLTs estimated the toxicity rate to be greater than 30% at any dose level, then the Executive Committee will be notified, and the committee would determine whether to stop accrual

2. Primary Outcome: Phase II: Overall Survival Rate at 2 Years (Including Phase I Patients at Same Dose)
Description: Survival time is defined as time from registration to date of death from any cause and is estimated by the Kaplan-Meier method. Patients last known to be alive are censored at the date of last contact. (Please note that this outcome measure is considered the primary endpoint for the Phase II component of the study, but that the patients from Phase I that were treated at the same dose level are included, as indicated in the treatment arm descriptions. )
Time Frame: Analysis occured after all patients have been on study for 2 years. Maximum follow-up at time of analysis was 8.5 years.
Population: Eligible patients on Temozolomide 100 mg arms who started study treatment
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Combined Temozolomide 100mg Arms: Phase I: Temozolomide 100mg and Phase II: Temozolomide 100 mg
Arm/Group | Combined Temozolomide 100mg Arms
Number analyzed (Participants) | 53
percentage of participants | 80.8 [70.1 to 91.5]
Statistical Analysis 1: Comparison: Combined Temozolomide 100mg Arms; Null hypothesis: Two-year survival rate <= 64%; Alternative hypothesis: Two-year survival rate > 64%. The fixed survival rate for comparison comes from Radiation Therapy Oncology Group (RTOG) trial 9310. (RTOG 9310 does not fall within ClinicalTrials.gov registration/reporting requirements.); Test type: Superiority; p = 0.006, One-sample z-test

3. Secondary Outcome: Phase II: Pre-irradiation Chemotherapy Tumor Response Rate (Including Phase I Patients at Same Dose)
Description: Tumor response was centrally reviewed. Complete response: Disappearance of all enhancing tumor, the patient must be off steroid therapy and neurologically stable or improved; partial response: ≥ 50% decrease in enhancing tumor; progressive disease: ≥ 25% increase in a lesion, progressive or newly emergent meningeal or ocular disease. (Please note that this outcome measure is considered a secondary endpoint for the Phase II component of the study, but that the patients from Phase I that were treated at the same dose level are included, as indicated in the treatment arm descriptions. )
Time Frame: From start of treatment to 10 weeks if RT received, to 15 weeks if not.
Population: Eligible patients on Temozolomide 100 mg arms who started study treatment and have scans for central review
Measure: Count of Participants; unit: Participants
Arm/Group | Combined Temozolomide 100mg Arms
Number analyzed (Participants) | 35
Participants
  Complete Response | 18
  Partial Response | 12
  Progressive Disease | 2
  Not evaluable | 3
Statistical Analysis 1: Comparison: Combined Temozolomide 100mg Arms; RTOG 93-10 reported a pre-irradiation chemotherapy complete response rate of 59%. A chi-square test with a 0.20 one-sided significance level provides 81% power to detect the difference between a null hypothesis complete response rate of 59% and the alternative rate of 71% (a 20% increase) for the planned sample size of 52 patients; Test type: Other; p = 0.82, Chi-squared; One-sample test of proportions

4. Secondary Outcome: Phase II: Progression-free Survival (Including Phase I Patients at Same Dose)
Description: Progression is defined as greater than 25% increase in enhancing tumor or the appearance of new lesions in the brain, eye, or the appearance of a new positive cerebrospinal fluid (CSF) cytology. The patient may be neurologically stable or worse and on stable or increasing doses of corticosteroid. Progression-free survival time is defined as time from registration to the date of progression, death, or last known follow-up (censored). Progression-free survival rates are estimated using the Kaplan-Meier method. (Please note that this outcome measure is considered a secondary endpoint for the Phase II component of the study, but that the patients from Phase I that were treated at the same dose level are included, as indicated in the treatment arm descriptions. )
Time Frame: Analysis occured after all patients have been on study for 2 years. Maximum follow-up at time of analysis was 8.5 years.
Population: Eligible patients on Temozolomide 100 mg arms who started study treatment
Measure: Median (95% Confidence Interval); unit: years
Arm/Group | Combined Temozolomide 100mg Arms
Number analyzed (Participants) | 53
years | 5.4 [1.8 to 7.3]

ADVERSE EVENTS:
Description: Subjects experiencing more than one of a given adverse event are counted only once for that adverse event.
Arm/Group | Phase I: Temozolomide 100 mg | Phase I: Temozolomide 150 mg | Phase II: Temozolomide 100 mg
Serious Adverse Events (participants affected / at risk) | 3/6 | 4/6 | 16/47
Other Adverse Events (participants affected / at risk) | 6/6 | 6/6 | 47/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase I: Temozolomide 100 mg (N=6) | Phase I: Temozolomide 150 mg (N=6) | Phase II: Temozolomide 100 mg (N=47)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Hemoglobin decreased (Blood and lymphatic system disorders) | 0 | 0 | 1
Vomiting NOS (Gastrointestinal disorders) | 0 | 0 | 1
Fatigue (General disorders) | 0 | 0 | 1
Late RT Toxicity:Other NOS (General disorders) | 0 | 0 | 1
Pain-other (General disorders) | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 0
Leukopenia NOS (Investigations) | 2 | 1 | 5
Neutropenia (Investigations) | 3 | 2 | 5
Platelet count decreased (Investigations) | 1 | 1 | 7
Alkalosis NOS (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyperglycemia NOS (Metabolism and nutrition disorders) | 0 | 0 | 2
Ataxia NEC (Nervous system disorders) | 0 | 0 | 1
Convulsions NOS (Nervous system disorders) | 0 | 1 | 0
Encephalopathy NOS (Nervous system disorders) | 0 | 0 | 1
Headache NOS (Nervous system disorders) | 0 | 0 | 1
Learning disorder NOS (Nervous system disorders) | 0 | 0 | 1
Peripheral motor neuropathy (Nervous system disorders) | 0 | 0 | 1
Speech disorder NEC (Nervous system disorders) | 0 | 0 | 2
Renal failure NOS (Renal and urinary disorders) | 1 | 0 | 0
Thrombosis NOS (Vascular disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phase I: Temozolomide 100 mg (N=6) | Phase I: Temozolomide 150 mg (N=6) | Phase II: Temozolomide 100 mg (N=47)
Hematologic-Other (Blood and lymphatic system disorders) | 0 | 1 | 2
Hemoglobin decreased (Blood and lymphatic system disorders) | 5 | 6 | 39
Hemolysis NOS (Blood and lymphatic system disorders) | 0 | 1 | 0
Platelet transfusion (Blood and lymphatic system disorders) | 2 | 0 | 3
Arrhythmia NOS (Cardiac disorders) | 0 | 1 | 2
Edema NOS (Cardiac disorders) | 3 | 2 | 12
Cushingoid (Endocrine disorders) | 1 | 0 | 1
Cataract NEC (Eye disorders) | 1 | 0 | 1
Diplopia (Eye disorders) | 0 | 1 | 5
Dry eye NEC (Eye disorders) | 1 | 0 | 3
Late RT Toxicity:Eye NOS (Eye disorders) | 2 | 0 | 5
Ocular-Other (Eye disorders) | 1 | 0 | 5
Vision blurred (Eye disorders) | 1 | 1 | 15
Constipation (Gastrointestinal disorders) | 3 | 1 | 11
Diarrhea NOS (Gastrointestinal disorders) | 1 | 2 | 11
Esophageal spasm (Gastrointestinal disorders) | 0 | 1 | 1
Esophagitis NOS (Gastrointestinal disorders) | 1 | 0 | 7
Nausea (Gastrointestinal disorders) | 5 | 4 | 32
Stomatitis (Gastrointestinal disorders) | 2 | 1 | 11
Vomiting NOS (Gastrointestinal disorders) | 5 | 1 | 25
Fatigue (General disorders) | 6 | 6 | 42
Late RT Toxicity:Other NOS (General disorders) | 2 | 1 | 10
Pain-other (General disorders) | 0 | 2 | 16
Rigors (General disorders) | 1 | 0 | 5
Hepatic-Other (Hepatobiliary disorders) | 2 | 1 | 2
Allergy-Other (Immune system disorders) | 3 | 0 | 0
Infection NOS (Infections and infestations) | 2 | 0 | 9
Infection with grade 3 or 4 neutropenia (Infections and infestations) | 0 | 1 | 5
Dermatitis radiation NOS (Injury, poisoning and procedural complications) | 3 | 3 | 17
Ecchymosis (Injury, poisoning and procedural complications) | 0 | 1 | 5
Late RT Toxicity:Skin(within RT field)NOS (Injury, poisoning and procedural complications) | 3 | 0 | 9
Operative injury of vein/artery (Injury, poisoning and procedural complications) | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 5 | 3 | 27
Aspartate aminotransferase increased (Investigations) | 4 | 2 | 24
Blood alkaline phosphatase NOS increased (Investigations) | 2 | 1 | 6
Blood bilirubin increased (Investigations) | 0 | 1 | 6
Blood creatinine increased (Investigations) | 3 | 1 | 15
Gamma-glutamyltransferase increased (Investigations) | 1 | 1 | 1
Leukopenia NOS (Investigations) | 4 | 5 | 26
Lymphopenia (Investigations) | 1 | 2 | 20
Metabolic-Other (Investigations) | 1 | 1 | 5
Neutropenia (Investigations) | 2 | 3 | 19
Platelet count decreased (Investigations) | 4 | 1 | 30
Prothrombin time prolonged (Investigations) | 0 | 1 | 2
Weight decreased (Investigations) | 2 | 3 | 10
Weight increased (Investigations) | 1 | 0 | 6
Anorexia (Metabolism and nutrition disorders) | 3 | 3 | 17
Blood albumin decreased (Metabolism and nutrition disorders) | 2 | 0 | 5
Blood bicarbonate decreased (Metabolism and nutrition disorders) | 1 | 0 | 1
Blood magnesium decreased (Metabolism and nutrition disorders) | 0 | 2 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 5
Hyperglycemia NOS (Metabolism and nutrition disorders) | 2 | 2 | 12
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 1 | 5
Hypernatremia (Metabolism and nutrition disorders) | 1 | 0 | 4
Hyperuricemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypocalcemia (Metabolism and nutrition disorders) | 5 | 4 | 26
Hypoglycaemia NOS (Metabolism and nutrition disorders) | 0 | 1 | 4
Hypokalemia (Metabolism and nutrition disorders) | 1 | 1 | 14
Hyponatremia (Metabolism and nutrition disorders) | 1 | 1 | 8
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 6
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Joint, muscle, or bone-Other (Musculoskeletal and connective tissue disorders) | 0 | 1 | 3
Muscle weakness NOS (Musculoskeletal and connective tissue disorders) | 2 | 1 | 10
Amnesia NEC (Nervous system disorders) | 2 | 2 | 14
Ataxia NEC (Nervous system disorders) | 2 | 2 | 13
Cerebral ischaemia (Nervous system disorders) | 1 | 0 | 0
Convulsions NOS (Nervous system disorders) | 0 | 1 | 5
Dizziness (exc vertigo) (Nervous system disorders) | 0 | 1 | 7
Headache NOS (Nervous system disorders) | 4 | 2 | 30
Late RT Toxicity:Brain NOS (Nervous system disorders) | 2 | 1 | 5
Late RT Toxicity:Encephalopathy NOS (Nervous system disorders) | 0 | 1 | 2
Neuralgia NOS (Nervous system disorders) | 0 | 1 | 7
Neurologic-Other (Nervous system disorders) | 1 | 1 | 3
Peripheral motor neuropathy (Nervous system disorders) | 3 | 3 | 15
Peripheral sensory neuropathy (Nervous system disorders) | 3 | 2 | 10
Speech disorder NEC (Nervous system disorders) | 3 | 0 | 6
Taste disturbance (Nervous system disorders) | 3 | 0 | 14
Tremor NEC (Nervous system disorders) | 1 | 0 | 0
Anxiety NEC (Psychiatric disorders) | 1 | 1 | 9
Confusion (Psychiatric disorders) | 0 | 1 | 9
Depression NEC (Psychiatric disorders) | 2 | 2 | 9
Insomnia NEC (Psychiatric disorders) | 2 | 0 | 10
Renal/GU-Other (Renal and urinary disorders) | 1 | 1 | 1
Urinary incontinence (Renal and urinary disorders) | 2 | 1 | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 6
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 4 | 2 | 24
Dermatitis exfoliative NOS (Skin and subcutaneous tissue disorders) | 1 | 1 | 11
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Pruritus NOS (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Skin-Other (Skin and subcutaneous tissue disorders) | 1 | 0 | 2
Hypertension NOS (Vascular disorders) | 3 | 0 | 6
Thrombosis NOS (Vascular disorders) | 1 | 0 | 5

LIMITATIONS AND CAVEATS:
The 200 mg/m^2 treatment arm in the phase I component of the study did not open. Outcome measures are categorized as the phase I or phase II study component, but phase I patients at corresponding dose level are included in the phase II analyses.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI's are required to abide by the sponsor's publication guidelines which require review by coauthors and subsequent review and approval by the sponsor.